CLINICAL TRIAL: NCT03859206
Title: A Comparative Study : Medical Thoracoscopy Versus Tube Thoracostomy in Early Management of Empyema .
Brief Title: Medical Thoracoscopy Versus Tube Thoracostomy in Management of Empyema .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, shahenda mohammed gamal el din, assistant lecturer , chest department and tuberculosis, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: medical thoracoscopy empyema
Record Dates: First submitted 2019-02-19; First posted 2019-03-01 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Empyema
Keywords: medical; Thoracoscopy; loculated; empyema
MeSH Terms: conditions — Empyema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- empyema patients having medical thoracoscopy (Experimental): patients having empyema will undergo medical thoracoscopy as follow :
  With the closed biopsy forceps, step by step, fibrinous septae will be perforated, the pleural space was irrigated with saline and fluid and fibrinopurulent material were aspirated and removed from the pleural cavity, the entire pleural cavity was inspected and biopsies were obtained from suspicious areas carefully by the biopsy forceps under vision. Multiple lesions were encountered, multiple biopsies were taken & If no lesion, biopsy from parietal pleura was obtained from any sites.
  the intervention : is breaking the septation within the loculated empyema
  Interventions: Other: Medical thoracoscopy
- tube thoracostomy in patients with empyema (No Intervention): after confirmation of diagnosis of empyema Following , a chest tube (gauge 26-28) will be introduced and connected to underwater seal. The wound was then closed around the tube by stitches to fix it in position.

INTERVENTIONS:
Other: Medical thoracoscopy — • With the closed biopsy forceps, step by step, fibrinous septae were perforated, the pleural space was irrigated with saline and fluid and fibrinopurulent material were aspirated and removed from the pleural cavity, the entire pleural cavity was inspected and biopsies were obtained from suspicious areas carefully by the biopsy forceps under vision. Multiple lesions were encountered, multiple biopsies were taken & If no lesion, biopsy from parietal pleura was obtained from any sites.
  Arms: empyema patients having medical thoracoscopy

SUMMARY:
Pleural empyema : is a collection of pus in the pleural cavity caused by microorganisms, usually bacteria.[1]

Medical thoracoscopy has played a marginal role in the treatment of empyema for a long time, but has become more and more established in recent years. It can be per-formed in analgo-sedation in a bronchoscopy suite. It is minimally invasive and costs are much lower compared to surgical VATS. The diagnostic and therapeutic power seems to be comparable to VATS, since several studies show success rates with medical thoracoscopy between 73 and 100% (2, 3) .

DETAILED DESCRIPTION:
Study Setting: Assuit university hospital - Chest department. endoscopy unit . the subjects will under go the following :

1. Thorough medical history .
2. Routine hematologic investigations .
3. Pleural fluid aspiration and analyses .

   .
4. Radiological investigation & Chest X ray and CT scan to localize pleural fluid collection and assess the echogenicity of the effusion. & Chest ultrasound. Loculated empyema defined as ultrasonographic presence of empyema loculations with presence of intrapleural septa.
5. Medical thoracoscopy (MT):

Medical thoracoscopy with single-port-of-entry technique will be performed in the bronchoscopy unit under local anesthesia and conscious sedation using midazolam (2 mg) or bethdein.

* To define the point of entry into the pleural cavity, an ultrasound will be carried out.
* vertical incision will be made with the scalpel (usually near the midaxillary line), through the skin and subcutaneous tissue, appropriate to the size of the trocar to be used, usually of approximately 10 mm, parallel with and in the middle of the selected intercostal space.
* Then the trocar will be inserted in a corkscrew motion until the sudden release of resistance (after passing the costal pleura) is felt, while holding the handle of the trocar firmly in the palm of the hand, as index finger is extended.
* Under direct vision with the thoracoscope, introduction of pneumothorax will be performed, and all pleural fluid will be removed, and the pleural cavity will be inspected.
* With the closed biopsy forceps, step by step, fibrinous septae were perforated, the pleural space was irrigated with saline and fluid and fibrinopurulent material were aspirated and removed from the pleural cavity, the entire pleural cavity was inspected and biopsies were obtained from suspicious areas carefully by the biopsy forceps under vision. Multiple lesions were encountered, multiple biopsies were taken & If no lesion, biopsy from parietal pleura was obtained from any sites.
* & Following thoracoscopy, a chest tube (gauge 26-28) was introduced and connected to underwater seal. The wound was then closed around the tube by stitches to fix it in position.
* & After the procedure, chest X- ray PA view was done to show if any complications had happened and to insure inflation of the lung, to determine the size of the residual pneumothorax.
* Vital signs were recorded at appropriate intervals for 24 h. & The rigid thoracoscope and its accessories were sterilized by cold immersion in 2% gultraldhyde (cidex) for at least 30 min.
* An intercostal drain will be placed with underwater seal drainage to drain residual air and fluid from the pleural cavity, allowing the lung to re expand.
* The indications for removal of chest tubes will be absence of air leakage and cessation of fluid flow (100-150 mL daily).

  * The patients who would be diagnosed will be blindly randomized to the two study arms :

medical thoracoscopy or tube thoracostomy .

ELIGIBILITY:
Inclusion Criteria:

1. unilateral or bilateral frank pleural empyema (pus) .
2. age > 18 and <70 years old

Exclusion Criteria:

1. Transudative pleural effusion.
2. Bleeding disorders.
3. Hemo-dynamically unstable patients.
4. General contraindications to thoracoscopy e.g. unstable angina, left ventricular failure, uncontrolled hypertension, bleeding tendency. . .etc.
5. Recent history of chest trauma or proved hemothorax.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Medical cure without secondary Intervention | up to 14 days .
  medical cure will be defined as radiologic confirmation of successful pleural drainage (i.e. reduction of the size of the pleural fluid on the chest X-ray and chest ultrasound )with no need for further treatment by r surgical interventions) objective evidence of sepsis resolution (improvement in temperature and clinical condition and decreasing inflammatory laboratory markers .and decrease of amount of fluid discharge less than (50-100)cc per day .

SECONDARY OUTCOMES:
Duration of hospital stay | up to 14 day .
  Reduction in hospital stay in group with medical thoracoscopy in comparison to the group with simple chest tube
Adverse events | within 24 hour after medical thoracoscopy
  such as bleeding , sever pain , persistence air leak

REFERENCES:
- [Background] Redden MD, Chin TY, van Driel ML. Surgical versus non-surgical management for pleural empyema. Cochrane Database Syst Rev. 2017 Mar 17;3(3):CD010651. doi: 10.1002/14651858.CD010651.pub2. PMID 28304084
- [Background] Brutsche MH, Tassi GF, Gyorik S, Gokcimen M, Renard C, Marchetti GP, Tschopp JM. Treatment of sonographically stratified multiloculated thoracic empyema by medical thoracoscopy. Chest. 2005 Nov;128(5):3303-9. doi: 10.1378/chest.128.5.3303. PMID 16304276